CLINICAL TRIAL: NCT02052141
Title: A Phase 3, Multicenter, Randomized, Single-Blind, Dose-Ranging, Crossover Study to Evaluate the Safety and Efficacy of Intravenous Administration of CINRYZE® (C1 Esterase Inhibitor [Human]) for the Prevention of Angioedema Attacks in Children 6 to 11 Years of Age With Hereditary Angioedema
Brief Title: Safety and Efficacy Study of CINRYZE for Prevention of Angioedema Attacks in Children Ages 6-11 With Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 0624-301; 2013-002453-29 (EudraCT Number); SHP616-301 (Other: Shire)
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Pediatric; C1 inhibitor; HAE; Cinryze; C1 INH; Prevention
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 500/1000 (Experimental): 500 Units of CINRYZE administered by IV injection twice per week for 12 weeks followed by 1000 Units of CINRYZE administered by IV injection twice per week for 12 weeks
  Interventions: Biological: CINRYZE 500; Biological: CINRYZE 1000
- 1000/500 (Experimental): 1000 Units of CINRYZE administered by IV injection twice per week for 12 weeks followed by 500 Units of CINRYZE administered by IV injection twice per week for 12 weeks
  Interventions: Biological: CINRYZE 500; Biological: CINRYZE 1000

INTERVENTIONS:
Biological: CINRYZE 500 — 500 Units of CINRYZE administered by IV injection
Biological: CINRYZE 1000 — 1000 Units of CINRYZE administered by IV injection

SUMMARY:
Primary Objective - To assess the relative efficacy of two dose levels of CINRYZE (500 Units and 1000 Units) administered by intravenous (IV) injection every 3 or 4 days to prevent angioedema attacks in children 6 to 11 years of age with hereditary angioedema (HAE).

Secondary Objectives - To assess the safety and tolerability, characterize the pharmacokinetics (PK) and pharmacodynamics (PD), and assess the immunogenicity of two dose levels of CINRYZE administered by IV injection in children 6 to 11 years of age with HAE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type I or Type II HAE.
* History of angioedema attacks.

Exclusion Criteria:

* History of bleeding or clotting abnormality.
* Diagnosis of acquired angioedema or known to have C1 INH antibodies.
* History of allergic reaction to C1 esterase inhibitor or other blood products.
* Receipt of any experimental agents other than those required for prevention or treatment of angioedema attacks within 30 days prior to screening.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- United States (3):
  - Asthma and Allergy Associates, P.C, Colorado Springs, Colorado
  - Nevada Access to Research and Education Society, Las Vegas, Nevada
  - Oregon Allergy Associates, Eugene, Oregon
- Germany (2):
  - Klinikum der J.W. Goethe Universitat, Frankfurt
  - HZRM Hamophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Instituto Nacional de Pediatria, Mexico City, Mexico
- Clinical County Hospital Mures, Târgu Mureş, Romania

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.shiretrials.com website. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Aygoren-Pursun E, Soteres D, Moldovan D, Christensen J, Van Leerberghe A, Hao J, Schranz J, Jacobson KW, Martinez-Saguer I. Preventing Hereditary Angioedema Attacks in Children Using Cinryze(R): Interim Efficacy and Safety Phase 3 Findings. Int Arch Allergy Immunol. 2017;173(2):114-119. doi: 10.1159/000477541. Epub 2017 Jun 30. PMID 28662509
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Aygoren-Pursun E, Soteres DF, Nieto-Martinez SA, Christensen J, Jacobson KW, Moldovan D, Van Leerberghe A, Tang Y, Lu P, Vardi M, Schranz J, Martinez-Saguer I. A randomized trial of human C1 inhibitor prophylaxis in children with hereditary angioedema. Pediatr Allergy Immunol. 2019 Aug;30(5):553-561. doi: 10.1111/pai.13060. Epub 2019 May 29. PMID 30968444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 10 study centers in the United States, European Union, Mexico, and Israel between 20 March 2014 (first participant first visit) and 04 May 2017 (last participant last visit).
Pre-assignment Details: A total of 16 participants were screened and of them, 12 were enrolled into the baseline observational period (12 weeks) and were randomized to receive the treatment in sequence A-B and B-A during this crossover study without a washout period.
Groups:
- Treatment A-B (500 U/1000 U CINRYZE): Participants received 500 units (U) of CINRYZE intravenous (IV) injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment A) during intervention period 1 followed by 1000 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment B) during intervention period 2. There was no washout period between the two intervention periods.
- Treatment B-A (1000 U/500 U CINRYZE): Participants received 1000 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment B) during intervention period 1 followed by 500 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment A) during intervention period 2. There was no washout period between the two intervention periods.
Period: Intervention Period 1
Arm/Group | Treatment A-B (500 U/1000 U CINRYZE) | Treatment B-A (1000 U/500 U CINRYZE)
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0
Period: Intervention Period 2
Arm/Group | Treatment A-B (500 U/1000 U CINRYZE) | Treatment B-A (1000 U/500 U CINRYZE)
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who took at least 1 dose of investigational product.
Groups:
- Treatment A-B (500 U/1000 U CINRYZE): Participants received 500 units (U) of CINRYZE intravenous (IV) injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment A) in Intervention period 1 followed by 1000 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment B) in Intervention period 2. There was no washout period between two intervention periods.
- Treatment B-A (1000 U/500 U CINRYZE): Participants received 1000 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment B) in Intervention period 1 followed by 500 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 12 weeks (Treatment A) in Intervention period 2. There was no washout period between two intervention periods.
- Total: Total of all reporting groups
Arm/Group | Treatment A-B (500 U/1000 U CINRYZE) | Treatment B-A (1000 U/500 U CINRYZE) | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age was calculated as the difference between date of birth and date of informed consent, truncated to years.
  Years | 10.2 (0.84) | 9.4 (1.51) | 9.8 (1.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Normalized Number of Angioedema Attacks Per Month in a Treatment Period
Description: Angioedema attack was defined as the participant-reported indication of symptoms or signs such as swelling or pain at any location following a report of no swelling or pain on the previous day. Manifestations of an attack that progress from one site to another, prior to complete resolution, was considered a single attack. Attacks that began to regress and then worsened before complete resolution was also considered one attack. Attacks that began then appeared to resolve and then reappeared without a symptom-free calendar day reported after the appearance of resolution were considered 1 attack. Any events of swelling due to trauma or symmetrical nonpainful swelling of the lower extremities were not considered an angioedema attack. The number of attacks was normalized for the number of days participants participated in a given period and expressed as the monthly frequency.
Time Frame: From start of treatment up to 12 weeks during each treatment period
Population: Full Analysis Set (FAS) included all participants in the safety set who had at least 1 post-baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: Angioedema attacks per month
Groups:
- Treatment A (500 U CINRYZE): Participants received 500 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 24 weeks (Intervention period 1 in sequence A-B and ntervention period 2 in sequence B-A). Each intervention period was of 12 weeks.
- Treatment B (1000 U CINRYZE): Participants received 1000 U CINRYZE IV injection twice weekly (every 3 or 4 days) for 24 weeks (Intervention period 2 in sequence A-B and ntervention period 1 in sequence B-A). Each intervention period was of 12 weeks.
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Angioedema attacks per month | 1.2 (1.53) | 0.7 (1.35)
Statistical Analysis 1: Comparison: Treatment A (500 U CINRYZE) vs Treatment B (1000 U CINRYZE); Test type: Superiority; p = 0.03, Paired t-test; Mean difference = -0.4, 90% CI 2-sided [-0.71 to -0.10], Standard Deviation 0.58 — The difference between treatment B over treatment A was estimated

2. Secondary Outcome: Cumulative Attack-severity Score of Angioedema Attacks Normalized Per Month in a Treatment Period
Description: Severity of the angioedema attack sign/symptom was characterized as None: no symptom; Mild: noticeable symptom but easily tolerated by the participant and did not interfere with routine activities; Moderate: symptom interfered with the participant's ability to attend school or participate in family life and social/recreational activities; Severe: symptom significantly limited the participant's ability to attend school or participate in family life and social/recreational activities. Symptom severity score was assigned as Mild = 1, Moderate = 2 and Severe = 3. Cumulative attack severity score was the sum of the maximum symptom severity scores recorded for each angioedema attack in a treatment period. Cumulative attack-severity score normalized per month [(raw score/number of days of participation in that treatment period)*30.4] was reported here. Cumulative attack-severity score normalized per month ranged from 0 to 10.4 and higher scores represent worse symptoms.
Time Frame: From start of treatment up to 12 weeks during each treatment period
Population: FAS included all participants in the safety set who had at least 1 post-baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Score on a scale | 2.0 (2.91) | 1.4 (2.68)
Statistical Analysis 1: Comparison: Treatment A (500 U CINRYZE) vs Treatment B (1000 U CINRYZE); Test type: Superiority; p = 0.05, Paired t-test; Mean difference = -0.7, 90% CI 2-sided [-1.20 to -0.11], Standard Deviation 1.06 — The difference between treatment B over treatment A was estimated

3. Secondary Outcome: Cumulative Daily-severity Score of Angioedema Attacks Normalized Per Month in a Treatment Period
Description: Severity of the angioedema attack sign/symptom was characterized as None: no symptom; Mild: noticeable but easily tolerated by the participant and did not interfere with routine activities; Moderate: interfered with the participant's ability to attend school or participate in family life and social/recreational activities; Severe: significantly limited the participant's ability to attend school or participate in family life and social/recreational activities. Symptom severity score was assigned as Mild = 1, Moderate = 2 and Severe = 3. Cumulative daily-severity score was the sum of the severity scores recorded for every day of reported symptoms in a treatment period. Cumulative daily-severity score normalized per month [(raw score/number of days of participation in that treatment period)*30.4] was reported here. Cumulative daily-severity score normalized per month ranged from 0 to 15.6 and higher scores represent worse symptoms.
Time Frame: From start of treatment up to 12 weeks during each intervention period
Population: FAS included all participants in the safety set who had at least 1 post-baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Score on a scale | 4.1 (5.01) | 2.2 (3.50)
Statistical Analysis 1: Comparison: Treatment A (500 U CINRYZE) vs Treatment B (1000 U CINRYZE); Test type: Superiority; p = 0.04, Paired t-test; Mean difference = -1.9, 90% CI 2-sided [-3.31 to -0.38], Standard Deviation 2.82 — The difference between treatment B over treatment A was estimated

4. Secondary Outcome: Normalized Number of Angioedema Attacks Per Month Requiring Acute Treatment in a Treatment Period
Description: Angioedema attack was defined as the participant-reported indication of symptoms or signs such as swelling or pain at any location following a report of no swelling or pain on the previous day. Manifestations of an attack that progress from one site to another, prior to complete resolution, was considered a single attack. Attacks that began to regress and then worsened before complete resolution was also considered one attack. Attacks that began then appeared to resolve and then reappeared without a symptom-free calendar day reported after the appearance of resolution were considered 1 attack. Any events of swelling due to trauma or symmetrical nonpainful swelling of the lower extremities were not considered an angioedema attack. The number of attacks requiring acute treatment was normalized for the number of days participants participated in a given period and expressed as the monthly frequency.
Time Frame: From start of treatment up to 12 weeks during each intervention period
Population: FAS included all participants in the safety set who had at least 1 post-baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: Angioedema attacks per month
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Angioedema attacks per month | 0.7 (1.5) | 0.4 (1.27)
Statistical Analysis 1: Comparison: Treatment A (500 U CINRYZE) vs Treatment B (1000 U CINRYZE); Test type: Superiority; p = 0.07, Paired t-test; Mean difference = -0.2, 90% CI 2-sided [-0.41 to -0.03], Standard Deviation 0.37 — The difference between treatment B over treatment A was estimated

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) by Dose Group
Description: An adverse event (AE) was any untoward, undesired, unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiological observations occurring in a participant participating in a clinical study with the sponsor's product, regardless of causal relationship. TEAEs were defined as events that started or worsened on or after the date and time of the first dose of investigational product and up to 7 days after the last dose of investigational product.
Time Frame: From start of study treatment up to 25 weeks
Population: Safety set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Participants | 10 | 11

6. Secondary Outcome: Plasma Concentration of C1 Esterase Inhibitor (C1 INH) Antigen
Description: C1 INH antigen concentration in plasma was determined using an automated nephelometric assay.
Time Frame: Pre-dose and 1 hour (h) post-dose at Week 1 (Dose 1) and Week 6 (Dose 12); Pre-dose, 1, 2, 4 and 8 h post-dose at Week 12 (Dose 24) of each intervention period
Population: Pharmacokinetic (PK) set consisted of all pariticipants in the safety set with no major deviations related to investigational product intake and evaluable PK profiles.
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Gram per liter (g/L)
  Week 1 (Pre-dose 1): number analyzed (Participants) | 12 | 11
  Week 1 (Pre-dose 1) | 0.0945 (0.03294) | 0.0736 (0.02885)
  Week 1 (1 h post-dose 1): number analyzed (Participants) | 11 | 11
  Week 1 (1 h post-dose 1) | 0.1819 (0.04331) | 0.2084 (0.08757)
  Week 6 (Pre-dose 12) | 0.0965 (0.03129) | 0.1068 (0.03098)
  Week 6 (1 h post-dose 12): number analyzed (Participants) | 10 | 11
  Week 6 (1 h post-dose 12) | 0.1631 (0.04188) | 0.2543 (0.05499)
  Week 12 (Pre-dose 24): number analyzed (Participants) | 12 | 11
  Week 12 (Pre-dose 24) | 0.0823 (0.02758) | 0.1002 (0.04420)
  Week 12 (1 h post-dose 24): number analyzed (Participants) | 12 | 10
  Week 12 (1 h post-dose 24) | 0.1621 (0.02990) | 0.2396 (0.04511)
  Week 12 (2 h post-dose 24): number analyzed (Participants) | 3 | 2
  Week 12 (2 h post-dose 24) | 0.1440 (0.00400) | 0.2070 (0.01838)
  Week 12 (4 h post-dose 24): number analyzed (Participants) | 2 | 2
  Week 12 (4 h post-dose 24) | 0.1440 (0.01131) | 0.1770 (0.02970)
  Week 12 (8 h post-dose 24): number analyzed (Participants) | 2 | 3
  Week 12 (8 h post-dose 24) | 0.1280 (0.00990) | 0.1790 (0.03100)

7. Secondary Outcome: C1 Esterase Inhibitor (C1 INH) Functional Activity in Plasma
Description: The functional activity of C1 INH in plasma samples was determined by a chromogenic assay.
Time Frame: Pre-dose and 1 h post-dose at Week 1 (Dose 1) and Week 6 (Dose 12); Pre-dose, 1, 2, 4 and 8 h post-dose at Week 12 (Dose 24) of each intervention period
Population: PK set consisted of all pariticipants in the safety set with no major deviations related to investigational product intake and evaluable PK profiles.
Measure: Mean (Standard Deviation); unit: Units per milliliter (U/mL)
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Units per milliliter (U/mL)
  Week 1 (Pre-dose 1): number analyzed (Participants) | 12 | 11
  Week 1 (Pre-dose 1) | 0.290 (0.0914) | 0.210 (0.1282)
  Week 1 (1 h post-dose 1): number analyzed (Participants) | 12 | 11
  Week 1 (1 h post-dose 1) | 0.575 (0.1358) | 0.725 (0.3100)
  Week 6 (Pre-dose 12) | 0.297 (0.1375) | 0.336 (0.0933)
  Week 6 (1 h post-dose 12): number analyzed (Participants) | 11 | 11
  Week 6 (1 h post-dose 12) | 0.570 (0.1190) | 0.865 (0.1550)
  Week 12 (Pre-dose 24): number analyzed (Participants) | 12 | 11
  Week 12 (Pre-dose 24) | 0.255 (0.1108) | 0.362 (0.1897)
  Week 12 (1 h post-dose 24): number analyzed (Participants) | 12 | 10
  Week 12 (1 h post-dose 24) | 0.531 (0.1330) | 0.803 (0.1906)
  Week 12 (2 h post-dose 24): number analyzed (Participants) | 3 | 3
  Week 12 (2 h post-dose 24) | 0.497 (0.0635) | 0.613 (0.2601)
  Week 12 (4 h post-dose 24): number analyzed (Participants) | 3 | 3
  Week 12 (4 h post-dose 24) | 0.497 (0.0058) | 0.590 (0.1803)
  Week 12 (8 h post-dose 24): number analyzed (Participants) | 3 | 3
  Week 12 (8 h post-dose 24) | 0.430 (0.0458) | 0.643 (0.0723)

8. Secondary Outcome: Plasma Concentration of Complement C4
Description: Concentration of Complement C4 in plasma was determined using an automated nephelometric assay.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Milligram per liter (mg/L)
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Milligram per liter (mg/L)
  Week 1 (Pre-dose 1): number analyzed (Participants) | 12 | 11
  Week 1 (Pre-dose 1) | 105.1 (39.38) | 71.2 (29.63)
  Week 1 (1 h post-dose 1): number analyzed (Participants) | 12 | 11
  Week 1 (1 h post-dose 1) | 99.7 (36.73) | 71.4 (33.20)
  Week 6 (Pre-dose 12) | 97.3 (37.26) | 121.3 (41.50)
  Week 6 (1 h post-dose 12): number analyzed (Participants) | 11 | 11
  Week 6 (1 h post-dose 12) | 88.0 (27.75) | 111.7 (41.75)
  Week 12 (Pre-dose 24): number analyzed (Participants) | 12 | 11
  Week 12 (Pre-dose 24) | 83.3 (21.63) | 111.6 (50.28)
  Week 12 (1 h post-dose 24): number analyzed (Participants) | 12 | 10
  Week 12 (1 h post-dose 24) | 79.2 (20.21) | 90.7 (27.72)
  Week 12 (2 h post-dose 24): number analyzed (Participants) | 3 | 3
  Week 12 (2 h post-dose 24) | 86.7 (4.93) | 94.3 (32.04)
  Week 12 (4 h post-dose 24): number analyzed (Participants) | 3 | 3
  Week 12 (4 h post-dose 24) | 89.3 (12.66) | 103.7 (32.35)
  Week 12 (8 h post-dose 24): number analyzed (Participants) | 3 | 3
  Week 12 (8 h post-dose 24) | 99.3 (11.02) | 114.7 (30.75)

9. Secondary Outcome: Number of Participants With C1 Esterase Inhibitor (C1 INH) Antibodies in Plasma
Description: The presence of C1 INH antibodies in plasma samples was determined using a proprietary enzyme-linked-immunosorbent-assay. Number of participants with C1 INH Antibodies was reported.
Time Frame: Pre-dose, 1 week post treatment (Week 13, Week 25) and 1 month post treatment follow-up (Week 28)
Population: Safety set included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 25
Arm/Group | Treatment A (500 U CINRYZE) | Treatment B (1000 U CINRYZE)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (500 U CINRYZE) (N=12) | Treatment B (1000 U CINRYZE) (N=12)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Vascular pain (Vascular disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (9) | 1 (9)
Infusion site pain (General disorders) | 1 (19) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 9 (41) | 8 (25)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (4)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 6 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-Traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (5)
Irritability (Psychiatric disorders) | 1 (7) | 1 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema marginatum (Skin and subcutaneous tissue disorders) | 2 (12) | 2 (12)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02052141/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT02052141/SAP_001.pdf